CLINICAL TRIAL: NCT04759170
Title: The Effects of Recorded Receptive Music Therapy on Oral Nutrition and the Well-being of the Italian Premature Baby: Prospective Randomized Controlled Study Mom, Dad and Music Therapist Singing Voice
Brief Title: The Effects of Recorded Receptive Music Therapy on Oral Nutrition and the Well-being of the Italian Premature Baby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Barbara Sgobbi, Music Therapist, Ospedale di Circolo - Fondazione Macchi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 186
Record Dates: First submitted 2021-01-28; First posted 2021-02-18 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Music Therapy
Keywords: Music therapy; Hrv; Premature; Preterm; Music recorded receptive; Parents voice; feeding time; music therapist voice
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mother Recorded Receptive Music Therapy Intervention (Other): The effects of recorded receptive music therapy on oral nutrition and the well-being of the Italian premature baby
  Interventions: Other: Music therapy
- Fother Recorded Receptive Music Therapy Intervention (Other): The effects of recorded receptive music therapy on oral nutrition and the well-being of the Italian premature baby
  Interventions: Other: Music therapy
- Music therapist Recorded Receptive Music therapy intervention (Other): The effects of recorded receptive music therapy on oral nutrition and the well-being of the Italian premature baby
  Interventions: Other: Music therapy
- No singing (Other): The effects of recorded receptive music therapy on oral nutrition and the well-being of the Italian premature baby
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — The effects of receptive music therapy on oral nutrition and the well-being of the Italian premature baby

SUMMARY:
The investigators have thought with a dedicated research group, to deepen the use of receptive music therapy so that it can improve the non-nutritive sucking of premature babies through listening to lullabies sung by parents and by the music therapist, which can reduce the use feeding tube and the negative effects on stress or growth of the newborn. The acquisition of oral skills and the achievement of a complete autonomous suction are of fundamental importance for the discharge of the preterm infant. Some studies published in the literature suggest that listening to the mother's voice and lullabies can represent a positive auditory stimulus for babies to support nutritional and non-nutritive sucking (NNS). Positive reinforcement is an effective development strategy for improving the feeding skills of preterm infants. A brief receptive music therapy intervention with the infant's personal pacifier that plays lullabies sung by both parents or by the music therapist could reduce the use of the feeding tube and the length of hospitalization. The possible negative effects of this stimulation on infant stress or growth remain to be explored. The aim of this study is not only to evaluate the benefits of positive reinforcement on the nutritional sucking competence of the premature baby, but at the same time also to observe the possible effects on his well-being and on his clinical stability.

DETAILED DESCRIPTION:
In preterm infant, oral feeding requires significant maturation of the nervous system to support coordination of the oropharyngeal muscles and breathing. Additionally, the energy expenditure required by nutritional sucking attempts further complicates the acquisition of oral feeding skills and must be balanced by caloric intake to achieve sufficient growth. Achievement of exclusive autonomous sucking typically occurs only between 34 and 36 post-conception weeks. However, delays in achieving full oral sucking are common and may prolong the infant's hospitalization.Non-nutritive sucking (NNS) is a coordinated motor skill that can be taught through an educational activity that conditions neuronal responses through positive reinforcement.The international literature demonstrates that, through a behavioral approach, the use of the pacifier during non-nutritive sucking promotes nutritional sucking in preterm infants, improving their attachment and bottle feeding, and determines the reduction of the length of stay in intensive care. and improved general well-being of the newborn.The use of receptive music therapy can therefore be supportive and represent a positive reinforcement for the development and acquisition of oral and nutritional skills of the preterm infant. By taking advantage of non-nutritive sucking it is possible to improve the suckling capacity of the newborn, his feeding speed, weight gain and consequently reduce the length of hospital stay. It is essential to achieve this result without negatively affecting the well-being and stability of the preterm infant.

Although musical studies in premature infants are limited, a 2014 study published in Pediatrics highlighted how music-specific and the maternal voice can positively reinforce the behavioral and neural responses of the preterm infant.On the other hand, the possible similar effects of reproduction, through the use of receptive music therapy of the song of the father and / or the music therapist, have not yet been investigated. The investigators therefore decided to design a prospective, randomized and controlled study to test the hypothesis that the parental (maternal and / or paternal) and / or music therapist's chant influences the well-being and / or stress of the newborn, evaluated through the parameter Heart Rate Variability (HRV), NNS development, nutritional sucking capacity, weight growth, and length of stay in premature infants compared to a control group of infants not subjected to sound stimulation . 40 premature babies will be recruited to be divided into 4 groups, after computerized randomization: n. 3 musical groups (mother song, father song, music therapist song) and 1 control group (not subjected to musical stimulation). Infants with gestational age at birth between the 23rd and 34th week of gestation will be included. Neonates with intraventricular hemorrhage (IVH) and periventricular leukomalacia (PVL) may also be enrolled. Only newborns in ventilatory support at the time of evaluation and newborns with maxillofacial malformations that may interfere with the ability to suck will be excluded from enrollment. Newborns will be evaluated when they reach 32 ° -34 ° post-conception weeks, the amount of milk taken orally (by sucking) must be less than 50% of the total enteral intake.Infants who have not passed the subsequent hearing screening test using AABR (Brain Stem Automatic Response Test) will be excluded from the analysis, which is expected to be performed after reaching the correct age limit.

OUTCOMES Positive reinforcement is an effective development strategy for improving the feeding skills of preterm infants. A short receptive music therapy intervention that reproduces lullabies sung by both parents or by the music therapist could positively influence the acquisition of nutritional skills and the growth of the preterm infant. Evaluating how this can affect the clinical stability of the newborn (and therefore on his state of stress, measured in terms of HRV) represents a fundamental and primary point to explore, in order to be able to make the possible use of receptive music therapy applicable in the strategy of positive reinforcement. The objective of this study is therefore to evaluate the tolerance of a receptive music therapy intervention (in terms of clinical stability, assessed through the HRV parameter) by the enrolled infants and to investigate any benefits of positive reinforcement obtained, through its use, on the acquisition of nutrition and growth skills of preterm infants.

Primary outcomes: clinical stability by measuring Heart Rate Variability (HRV)

• The primary objective of this study is to evaluate and monitor the tolerance of receptive music therapy (in terms of measurement of the clinical stability parameter HRV) by infants during music therapy treatment.

Secondary outcomes: effects of positive reinforcement (carried out through the use of receptive music therapy) on the acquisition of food skills and the growth of preterm infants. In particular:

* Evaluation of the achievement of exclusive oral sucking (determined as a week post-conception and / or days of life).
* Evaluation of the variation in the speed of meal intake between the beginning and the end of the intervention (measured as the volume of the nutritional intake in milliliters divided by the time in minutes required for consumption).
* Evaluation of the weight gain of the newborn in the 24 hours following stimulation
* (expressed as a percentage of weight gain from enrollment).
* Assessment of the growth rate from the last day of treatment to discharge.
* Length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age at birth between the 23rd and 34th week of gestation
* Neonates with intraventricular hemorrhage (IVH)
* Neonates with periventricular leukomalacia (PVL)

Exclusion Criteria:

* Only newborns in ventilatory support at the time of evaluation
* Newborns with maxillofacial malformations
* Newborns will be evaluated when they reach 32 ° -34 ° post-conception weeks, the amount of milk taken orally (by sucking) must be less than 50% of the total enteral intake
* Infants who have not passed the next hearing screening test using AABR (Brain Stem Automatic Response Test), which is expected to be performed after reaching the correct age term

Ages: 23 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Clinical stability by measuring Heart Rate Variability (HRV) | 8 day
  Evaluate and monitor the tolerance of recorded receptive music therapy on clinical stability parameter HRV

SECONDARY OUTCOMES:
Effects of positive reinforcement carried out through the use of recorded receptive music therapy | through study completion, an average of 20 weeks
  Evaluation of the achievement of exclusive oral sucking
Effects of recorded receptive music therapy on positive reinforcement on the acquisition of food skills | through study completion, an average of 20 weeks
  Evaluation of the variation in the speed of meal intake between the beginning and the end of the intervention.
Effects of the use of recorded receptive music therapy on the acquisition in skill of preterm infants. | through study completion, an average of 20 weeks
  Evaluation of the weight gain of the newborn in the 24 hours following stimulation.
Effects of positive reinforcement carried out through the use of recorded receptive music therapy on the acquisition of food the growth of preterm infants. | through study completion, an average of 20 weeks
  Assessment of the growth rate from the last day of treatment to discharge.

OTHER OUTCOMES:
Length of hospital stay after music therapy treatment | through study completion, an average of 20 weeks
  Length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Agosti, MD, Principal Investigator — Neonatologia, TIN e Pediatria Verbano- Ospedale F. del Ponte
Locations (1):
- Ospedale F. Del Ponte, Varese, Italy

IPD SHARING:
Plan to Share IPD: No